CLINICAL TRIAL: NCT01331590
Title: A Pilot Study of G-CSF to Disrupt the Bone Marrow Microenvironment in Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Disrupting the Bone Marrow Microenvironment With G-CSF in Acute Lymphoblastic Leukemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201104323
Record Dates: First submitted 2011-03-31; First posted 2011-04-08 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Ifosfamide; Etoposide; etoposide phosphate; Dexamethasone; Calcium Dobesilate; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-CSF + Ifosfamide + Etoposide + Dexamethasone + Mesna (Experimental): G-CSF = 10 mcg/kg/d SQ starting on day 1 and continuing until ANC >=1000/mcL x 2 days
  Ifosfamide = 3330 mg/m2/d CIVI over 24 hours on Days 4-6
  Etoposide = 150 mg/m2 IV over 2 hours BID on Days 4-6
  Dexamethasone = 5 mg/m2 PO or IV BID on Days 4-10
  Mesna = 2660 mg/m2/d continuous IV infusion over 24 hours on Days 4-6. 2000 mg/m2 continuous IV infusion over 12 hours on Day 7 to be started immediately after completion of ifosfamide.
  Interventions: Drug: G-CSF; Drug: Ifosfamide; Drug: Etoposide; Drug: Dexamethasone; Drug: Mesna

INTERVENTIONS:
Drug: G-CSF
  Other Names: Filgrastim; Neupogen; Granulocyte Colony-Stimulating Factor; Recombinant Methionyl Human G-CSF
Drug: Ifosfamide
  Other Names: Ifex; Isophosphamide
Drug: Etoposide
  Other Names: Etopophos; VP-16
Drug: Dexamethasone
  Other Names: Decadron
Drug: Mesna
  Other Names: Mesnex

SUMMARY:
The purpose of this study is to determine the ability of G-CSF to disrupt the bone marrow microenvironment as a means to increase the efficacy of chemotherapy in patients with relapsed or refractory acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
In this study, we will combine G-CSF as priming prior to and during the administration of salvage chemotherapy regimen in ALL. Abundant data suggests that leukemic cells receive key growth and survival signals from the bone marrow microenvironment. Our preclinical data show that 4-5 days of G-CSF treatment is associated with a loss of osteoblasts and decreases expression of key chemokine/ cytokines which support lymphocyte development. The investigators hypothesize that G-CSF will disrupt the protective effects of the bone marrow microenvironment and augment the effect of chemotherapy in adults with ALL. This is a pilot study of G-CSF priming in adult patients with relapsed or refractory ALL to determine the feasibility and to characterize the effect of G-CSF treatment on the marrow microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia diagnosed according to WHO criteria (>25% lymphoblasts in BM) which is relapsed or refractory to therapy. Patients with t(9;22) must be refractory to BCR-ABL tyrosine kinase inhibitors.
* Age ≥ 18 years
* ECOG performance status ≤ 3.
* Adequate organ function defined as:

  * Calculated creatinine clearance ≥ 50 ml/min
  * AST, ALT, total bilirubin ≤ 2 x institutional ULN except when in the opinion of treating physician elevated levels are due to direct involvement of leukemia (eg. hepatic infiltration or biliary obstruction due to leukemia)
* Women of childbearing potential and sexually active males must be willing and able to use effective contraception while on study.
* Able to provide signed informed consent prior to registration on study.

Exclusion Criteria:

* Previous salvage chemotherapy with ifosfamide and etoposide
* Pregnant or nursing
* Received any other investigational agent or cytotoxic chemotherapy within the preceding 2 weeks
* Received colony stimulating factors filgrastim or sargramostim within 1 week or pegfilgrastim within 2 weeks of study
* Severe concurrent illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality | 30 days after start of treatment
Delayed hematologic recovery | Day 46 of treatment
  Defined as neutrophil recovery (ANC > 1,000/mm3) > 42 days after the start of chemotherapy in the absence of persistent leukemia

SECONDARY OUTCOMES:
Complete remission rate cytogenetic complete remission | 42 days
Overall survival | 2 years
  Every 6 months
Disease-free survival | 2 years
  Every 6 months
Remission duration | 2 years
  Every 6 months
Frequency and severity of adverse events | 30 days post treatment
Interaction of pretreatment disease and patient characteristics on clinical outcomes | Baseline
  Morphology, cytogenetics, immunophenotype, WBC, and performance status

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Uy, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu